CLINICAL TRIAL: NCT02379676
Title: Comparison of the Effects of Ticagrelor Versus Clopidogrel on Endothelial Dysfunction and Vascular Inflammation in Patients With Prior Non-ST-segment Acute Coronary Syndrome
Brief Title: Effect of Ticagrelor Versus Clopidogrel on Endothelial Dysfunction and Vascular Inflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kiyuk Chang (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Kiyuk Chang, Chief of the divison of cardiology, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC14MIMI0092k
Record Dates: First submitted 2015-02-28; First posted 2015-03-05 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Endothelial Dysfunction; Vascular Inflammation
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90mg twice daily
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel 75mg once daily
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90mg twice daily for 30 days
  Arms: Ticagrelor
Drug: Clopidogrel — Clopidogrel 75mg once daily for 30 days
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to compare the effects of ticagrelor and clopidogrel on endothelial dysfunction and vascular inflammation

Ticagrelor will lead to beneficial pleiotropic effects compared with treatment with clopidogrel in patients receiving a drug-eluting stents (DES) during percutaneous coronary intervention (PCI) for non-ST-segment acute coronary syndrome (NSTE-ACS) beyond 1 month after the index event. Ticagrelor treatment will improve percent flow-mediated dilation (FMD) values and reduces inflammatory gene expression on peripheral blood mononuclear cells.

DETAILED DESCRIPTION:
The primary objective of this study lies in whether ticagrelor improves endothelial dysfunction compared to clopidogrel, measured by endothelium-dependent flow-mediated dilation (FMD). The secondary objective is to demonstrate whether ticagrelor has an anti-atherosclerotic effect compared to clopidogrel in terms of reducing systemic low-grade inflammation. Endpoints are 1) difference of flow-mediated dilation values, and 2) messenger ribonucleic acid (mRNA) expression measured by quantitative real-time reverse transcription-polymerase chain reaction (qRT-PCR) of inflammation-associated key genes in circulation monocytes between non-ST-segment acute coronary syndrome patients treated with ticagrelor and clopidogrel.

Patients who agree to participate study are screened at Visit 1 (30 ~ 365 days after index percutaneous coronary intervention). Patients with endothelial dysfunction defined as screening flow-mediated dilation are randomly assigned at Visit 2 (0~7 days after screening test). And then, patients should receive study drugs according to allocated groups from the day of randomization. Ticagrelor 90mg twice daily or clopidogrel 75mg daily will be maintained for 30 days. Flow-mediated dilation are performed at screening and at Visit 3 (day 30 from the treatment of study drugs) and blood sampling are performed before the first dose of study drugs at Visit 2 and at Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Men and women ≥20 years of age
* Documented history of non-ST-segment acute coronary syndrome occurring 30 ~ 365 days prior to randomization and successfully treated with percutaneous coronary intervention using drug-eluting stent
* Patient currently prescribed and tolerating aspirin 100mg and clopidogrel 75mg.
* Patient who have demonstrated endothelial dysfunction defined as percent flow-mediated dilation values lower than 7% at baselines test

Exclusion Criteria:

* Patients with angina related symptoms
* Patients who did not undergo or failed invasive treatment
* Patients with a history of hypersensitivity to ticagrelor or clopidogrel
* Patients who took an anti-coagulant, anti-thrombotic regularly before the study, or plan to have continuous treatment during the study
* Patients who took vasoactive agents or caffeine ingestion for <48
* Patients with decompensated congestive heart failure of cardiogenic shock (Killip classification III or IV)
* Patients with intractable arrhythmia
* Patients with intractable arrhythmia
* Patients with second or third degree atrioventricular block
* Patients with uncontrolled hypertension
* Patients with high risk of hemorrhage like blood coagulation disorders, gastrointestinal bleeding, gross hematuria, intraocular bleeding, hemorrhagic stroke, intracranial hemorrhage
* Patients with more than moderate chronic obstructive pulmonary disease diagnosed by symptoms or documented by pulmonary function test
* Patients who required renal replacement therapy
* Patients with moderate to severe hepatic impairment
* Patients with platelet <100,000/μL
* Patients with hematocrit <30%
* Concomitant oral or parenteral therapy with strong cytochrome P450 3A4 inhibitors, cytochrome P450 3A substrates with narrow therapeutic indices, or strong cytochrome P450 3A4 inducers i) Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (but not erythromycin or azithromycin), nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir, over 1 litre daily of grapefruit juice ii) Substrates with narrow therapeutic index: cyclosporine, quinidine, simvastatin at doses >40 mg daily or lovastatin at doses >40 mg daily iii) Strong inducers: rifampin/rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital
* Patient who need to take drugs other than study medications and allowed concomitant medications during study period.
* Patients who have planned elective surgery or invasive procedure requiring temporary discontinued study medication during study period.
* Patients who are pregnant, breast feeding and not using medically acceptable birth control.
* Patients considered as unsuitable based on medical judgment by investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in percent flow-mediated dilation (FMD) values | Baseline, 30 days

SECONDARY OUTCOMES:
Percent flow-mediated dilation (FMD) values | Baseline, 30 days
Incidence rate of patient with percent flow-mediated dilation (FMD) value less than 7% | Baseline, 30 days
Inflammatory gene expression levels by quantitative real-time reverse transcription-polymerase chain reaction (qRT-PCR) | Baseline, 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, The Catholic.University of Korea
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea